CLINICAL TRIAL: NCT05947591
Title: Influence of Gait and Running on Foot Posture Index and Navicular Drop Modifications for Non-athletes.
Brief Title: Influence of Gait and Running on Foot Posture
Status: Completed | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, PhD, University of Seville
Other Study IDs: 0973-N-20
Record Dates: First submitted 2023-06-28; First posted 2023-07-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Foot Pronation in Healthy Adult
Keywords: run; pronation; adult; sport

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: healthy adults than gait over 1 hour,
  Interventions: Behavioral: foot posture index
- experimental: healthy adults that run over 1 hour
  Interventions: Behavioral: foot posture index

INTERVENTIONS:
Behavioral: foot posture index — the tendency to foot pronation in healthy subjects will be compared during one hour of walking versus one hour of running in subjects who usually run.
  Other Names: Navicular drop test

SUMMARY:
Objective: To evaluate in a sample of healthy non-athlete subjects, if the foot tends to a pronated position during a period of running compared to walking, evaluated during and after one hour after performing said activity.

Design: Quasi-experimental study, experimental and control group. Setting: Subjects who attend the Podiatry Clinical Area of the University of Seville.

Participants: N=72 healthy non-athlete volunteer adults who regularly run.

DETAILED DESCRIPTION:
Interventions: The volunteers will participate in the research on three occasions, the day of data collection, one day when they will carry out a one-hour walking period and on another occasion where they will carry out an hour of running. Changes in foot posture [FPI] or foot pronation position (navicular drop [ND]) were identified in various periods of time at the time of the initial assessment and examination (p1), after 30 minutes of walking or running ( p2), 45 minutes of walking or running (p3) and 60 minutes of walking or running (p4) of the activity elapsed.

Main outcome measures: Foot position will be measured using the Foot Posture Index (FPI) and navicular height using the navicular drop test (ND) at p1, p2, p3 and p4.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are: healthy adults, of both sexes, who come to the center on the indicated date and who are professional athletes but who do practice some regular physical activity, understood as running for one hour three times a week as minimum.

-

Exclusion Criteria:

a congenital or traumatic foot deformity, wearing plantar supports, pregnancy or being in current rehabilitation treatment or serious illness.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy non atletes subjects
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Foot posture index | 15 minutes
  The FPI consists of 6 criteria obtained from the subject's foot where each of them gives a score from -2 to +12. Its use is simple and is scientifically validated.
  The subject must be in a comfortable standing position where they support their feet as they usually do naturally. Its realization lasts approximately 2 minutes maximum for each of the feet, and after its execution an independent total value is obtained for each one of them that indicates a pronated, supinated or normal posture that goes from -12 to +12 value. .
navicular drop test | 15 minutes
  to evaluate the difference between the original height of the navicular tuberosity in sitting position and in load corresponds to the drop of the scaphoids, therefore, to the descent of the internal longitudinal arch

SECONDARY OUTCOMES:
Foot posture index | 60 minutes
  The FPI consists of 6 criteria obtained from the subject's foot where each of them gives a score from -2 to +12. Its use is simple and is scientifically validated.
  The subject must be in a comfortable standing position where they support their feet as they usually do naturally. Its realization lasts approximately 2 minutes maximum for each of the feet, and after its execution an independent total value is obtained for each one of them that indicates a pronated, supinated or normal posture that goes from -12 to +12 value. .
Navicular drop test | 60 minutes
  o evaluate the difference between the original height of the navicular tuberosity in sitting position and in load corresponds to the drop of the scaphoids, therefore, to the descent of the internal longitudinal arch

CONTACTS AND LOCATIONS:
Locations (1):
- Aurora Castro Mendez, Seville, Spain

IPD SHARING:
Plan to Share IPD: No